CLINICAL TRIAL: NCT05430854
Title: An Open-Label Extension Study To Evaluate The Long- Term Safety And Tolerability Of Daxdilimab (Hzn-7734) In Subjects With Systemic Lupus Erythematosus
Brief Title: Study of Daxdilimab (HZN-7734) for the Treatment of Systemic Lupus Erythematosus in an Open-label Extension Study
Acronym: RECAST SLE OLE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZNP-DAX-204
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Daxdilimab (Experimental): Daxdilimab injections over a total of 48 weeks.
  Interventions: Biological: Daxdilimab

INTERVENTIONS:
Biological: Daxdilimab — Daxdilimab will be administered subcutaneously as two injections for each dose.
  Other Names: HZN-7734

SUMMARY:
A Phase 2, Open-Label Extension study to evaluate the long-term safety and tolerability of daxdilimab in participants with Systemic Lupus Erythematosus completing the treatment period of the RECAST SLE clinical study.

DETAILED DESCRIPTION:
Approximately 156 participants will be enrolled to receive daxdilimab administered subcutaneously over 48 weeks. The maximum trial duration per participant is approximately 56 weeks, including the 48 weeks for the open-label treatment period where participants will receive daxdilimab and approximately 8 weeks for the follow-up period. Safety evaluations will be performed regularly throughout the course of the study.

Acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to understand and provide written informed consent.
* Must have completed the treatment period in the RECAST SLE study.
* Women of childbearing potential must have a negative urine pregnancy test on Day 1.
* Nonsterilized male subjects who are sexually active with a woman partner of childbearing potential must agree to use a condom with spermicide from Day 1 and until 3 months (approximately 5 half-lives) after receipt of the last dose.

Exclusion Criteria:

* Any condition or change during the RECAST SLE study that in the opinion of the Investigator or the Sponsor would interfere with evaluation and interpretation of subject safety or alter the risk-benefit associated with IP administration.
* Participation in another clinical study with an IP during the RECAST SLE study period.
* Planned elective surgeries that in the opinion of the Investigator or the Sponsor would interfere with evaluation and interpretation of subject safety.
* Any herpes zoster, cytomegalovirus, or Epstein-Barr virus infection that was not completely resolved prior to Visit 1.
* Clinically significant active infection at Visit 1, in the opinion of the Investigator.
* Pregnant or lactating females.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (52):
- United States (14):
  - Inland Rheumatology Clinical Trials Incorporated, Upland, California
  - Clinical Research of West Florida Inc - Clearwater, Clearwater, Florida
  - Millennium Research, Ormond Beach, Florida
  - IRIS Research and Development LLC, Plantation, Florida
  - Clinical Research of West Florida Inc - Tampa, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Bluegrass Community Research Inc, Lexington, Kentucky
  - NYU Langone Ambulatory Care Brooklyn Heights, Brooklyn, New York
  - DJL Clinical Research, Charlotte, North Carolina
  - Paramount Medical Research and Consulting LLC, Middleburg Heights, Ohio
  - Precision Comprehensive Clinical Research Solutions, Colleyville, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Southwest Rheumatology Research, LLC, Mesquite, Texas
  - Spectrum Medical, Inc, Danville, Virginia
- Argentina (7):
  - Consultorios Médicos Dr. Doreski, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Clínica Adventista Belgrano, Estomba, Buenos Aires
  - Framingham Centro Médico, La Plata, Buenos Aires
  - Instituto CER S.A, Quilmes, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes SRL, Quilmes, Buenos Aires
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Consultorio de Investigaciones Reumatologicas, San Miguel de Tucumán, Tucumán Province
- Greece (4):
  - Athens General Hospital 'G Gennimatas, Athens
  - Laiko General Hospital of Athens, Athens
  - University General Hospital of Larissa, Larissa
  - Kianous Stavros, Thessaloniki
- India (5):
  - Krishna Institute of Medical Sciences, Secunderabad, Andhra Pradesh
  - AES - AS - Panchshil Hospital - Ahmedabad, Ahmedabad, Gujarat
  - AES - AS - Unity Trauma Center and ICU - Unity Hospital - Surat, Surat, Gujarat
  - AES - AS - Sushruta Multispeciality Hospital & Research Center Pvt Ltd - Hubli, Hubli, Karnataka
  - Jasleen Hospital, Nagpur, Maharashtra
- Mexico (9):
  - Centro de Investigación en Artritis y Osteoporosis, Mexicali, Estado de Baja California
  - Morales Vargas Centro de Investigacion SC, León, Guanajuato
  - Bioclinica - Centro Integral En Reumatologia Sociedad Anónima de Capital Variable, Guadalajara, Jalisco
  - Investigacion Biomedica para el Desarrollo de Farmacos S.A. de C.V., Zapopan, Jalisco
  - Centro de Investigación y Tratamiento Reumatológico S.C, San Miguel, Mexico City
  - Centro Peninsular de Investigacion S.C.P, Mérida, Yucatán
  - Clinica de Investigacion en Reumatologia y Obesidad, Guadalajara
  - Centro de Estudios de Investigacion Basica Y Clinica SC, Jalisco
  - Consultorio de Reumatologia, Mexico City
- Poland (8):
  - Klinika Reumatologii i Rehabilitacji Ortopedyczno-Rehabilitacyjny Szpital Kliniczny im W. Degi, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne Plejady, Krakow, Lesser Poland Voivodeship
  - Pratia MCM, Krakow, Lesser Poland Voivodeship
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól, Lubusz Voivodeship
  - Medycyna Kliniczna Marzena Waszczak-Jeka, Warsaw, Masovian Voivodeship
  - Centrum Medyczne AMED, Warsaw, Masovian Voivodeship
  - Nasz Lekarz Osrodek Badan Klinicznych, Bydgoszcz
  - Centrym Medyczne AMED oddzial w Lodzi, Lodz, Łódź Voivodeship
- Serbia (3):
  - Institute of Rheumatology Belgrade, Belgrade
  - Military Medical Academy, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
- Hospital Universitario A Coruña, A Coruña, Spain
- National Taiwan University Hospital, Taipei, Province of China, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label extension (OLE) of study VIB7734.P2.S1 (NCT04925934). Eligible participants were enrolled after the completion of the VIB7734.P2.S1 study. 155 participants were enrolled at 54 centers in the United States, Argentina, Greece, India, Mexico, Poland, Serbia, Spain and Taiwan from 01 June 2022 to 31 October 2023.
Groups:
- Placebo/Daxdilimab 200 mg Every 12 Weeks (Q12W): Participants who received placebo in the parent study received daxdilimab 200 mg subcutaneous (SC) injection Q12W in this OLE Study.
- Daxdilimab 200 mg Every 4 Weeks (Q4W)/Daxdilimab 200 mg Q12W: Participants who received 200 mg Q4W in the parent study received daxdilimab 200 mg SC injection Q12W in this OLE Study.
- Daxdilimab 200 mg Q12W/Daxdilimab 200 mg Q12W: Participants who received 200 mg Q12W in the parent study received daxdilimab 200 mg SC injection Q12W in this OLE Study.
Period: Overall Study
Arm/Group | Placebo/Daxdilimab 200 mg Every 12 Weeks (Q12W) | Daxdilimab 200 mg Every 4 Weeks (Q4W)/Daxdilimab 200 mg Q12W | Daxdilimab 200 mg Q12W/Daxdilimab 200 mg Q12W
Started | 47 | 57 | 51
Completed | 8 | 4 | 5
Not Completed | 39 | 53 | 46
Not completed — Trial terminated by Sponsor | 39 | 50 | 46
Not completed — Withdrawal by Subject | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: OLE Safety Analysis Set: all participants who received at least 1 dose of daxdilimab in the OLE study.
Groups:
- Placebo/Daxdilimab 200 mg Q12W: Participants who received placebo in the parent study received daxdilimab 200 mg SC injection Q12W in this OLE Study.
- Daxdilimab 200 mg Q4W in Parent Study: Participants who received 200 mg Q4W in the parent study received daxdilimab 200 mg SC injection Q12W in this OLE Study.
- Total: Total of all reporting groups
Arm/Group | Placebo/Daxdilimab 200 mg Q12W | Daxdilimab 200 mg Q4W in Parent Study | Daxdilimab 200 mg Q12W/Daxdilimab 200 mg Q12W | Total
Number analyzed (Participants) | 47 | 57 | 51 | 155
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.3 (10.3) | 44.8 (12.8) | 45.9 (11.2) | 44.1 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 52 | 46 | 142
  Male | 3 | 5 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 24 | 16 | 59
  Not Hispanic or Latino | 28 | 33 | 35 | 96
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 1 | 2 | 0 | 3
  Asian | 7 | 5 | 8 | 20
  Black or African American | 3 | 5 | 6 | 14
  White | 35 | 39 | 35 | 109
  Other | 1 | 6 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of an IP, whether or not considered related to the IP. A TEAE is defined as any AE with an onset date on or after the first dose date in the OLE study.
Time Frame: Up to approximately 56 weeks
Population: OLE Safety Analysis Set: all participants who received at least 1 dose of daxdilimab in the OLE study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Daxdilimab 200 mg Q12W | Daxdilimab 200 mg Q4W in Parent Study | Daxdilimab 200 mg Q12W/Daxdilimab 200 mg Q12W
Number analyzed (Participants) | 47 | 57 | 51
Participants | 25 | 31 | 31

2. Primary Outcome: Number of Participants Who Experienced Serious Adverse Events (SAEs)
Description: An AE is considered "serious" if, in the view of either the Investigator or Sponsor, it results in any of the following outcomes:
  * Death
  * A life-threatening AE
  * Inpatient hospitalization or prolongation of existing hospitalization
  * Persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions
  * A congenital abnormality/birth defect
  * Important medical events judged to jeopardize the participant(s).
Time Frame: Up to approximately 56 weeks
Population: OLE Safety Analysis Set: all participants who received at least 1 dose of daxdilimab in the OLE study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Daxdilimab 200 mg Q12W | Daxdilimab 200 mg Q4W in Parent Study | Daxdilimab 200 mg Q12W/Daxdilimab 200 mg Q12W
Number analyzed (Participants) | 47 | 57 | 51
Participants | 3 | 5 | 5

3. Primary Outcome: Number of Participants Who Experienced AEs of Special Interest (AESI)
Description: An AESI is an AE of scientific and medical interest specific to understanding of the IP and may require close monitoring and collection of additional information by the Investigator. In this study, AESIs were:
  * Hypersensitivity reaction, including anaphylaxis
  * Severe (Grade 3 or higher) viral infections/reactivations
  * Opportunistic infections
  * Malignancy (except non-melanoma skin cancer).
Time Frame: Up to approximately 56 weeks
Population: OLE Safety Analysis Set: all participants who received at least 1 dose of daxdilimab in the OLE study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Daxdilimab 200 mg Q12W | Daxdilimab 200 mg Q4W in Parent Study | Daxdilimab 200 mg Q12W/Daxdilimab 200 mg Q12W
Number analyzed (Participants) | 47 | 57 | 51
Participants | 1 | 2 | 1

4. Secondary Outcome: Serum Concentration of Daxdilimab
Description: Serum concentration of daxdilimab refers to the amount of daxdilimab present in the blood serum at a given time. Blood samples were collected via venipuncture at the specified time frames. Week 0 corresponds to the last day of the treatment period in the parent study and Day 1 of the treatment period in the OLE study.
Time Frame: Week 0 (Week 0 = Day 1), Week 12, Week 24, Week 36, Week 48, Week 56
Population: PK Analysis Set: all participants who received any dose of daxdilimab in OLE study and had at least 1 measurable PK concentration post dose. Number analyzed represents the number of participants with available data at that time point.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Placebo/Daxdilimab 200 mg Q12W | Daxdilimab 200 mg Q4W in Parent Study | Daxdilimab 200 mg Q12W/Daxdilimab 200 mg Q12W
Number analyzed (Participants) | 47 | 57 | 51
ug/mL
  Week 0: number analyzed (Participants) | 0 | 55 | 50
  Week 0 |  | 5.527 (4.412) | 0.458 (0.614)
  Week 12 | 0.291 (0.390) | 0.502 (0.740) | 0.400 (0.520)
  Week 24: number analyzed (Participants) | 47 | 56 | 50
  Week 24 | 0.414 (0.575) | 0.398 (0.531) | 0.437 (0.437)
  Week 36: number analyzed (Participants) | 27 | 26 | 25
  Week 36 | 0.508 (0.616) | 0.464 (0.467) | 1.002 (1.404)
  Week 48: number analyzed (Participants) | 11 | 10 | 11
  Week 48 | 0.813 (1.044) | 0.380 (0.395) | 0.815 (0.759)
  Week 56: number analyzed (Participants) | 5 | 2 | 5
  Week 56 | 0.399 (0.251) | 0.146 (0.009) | 0.997 (0.898)

5. Secondary Outcome: Change From Baseline in Plasmacytoid Dendritic Cell (pDCs) Count
Description: PDCs count refers to the number of pDCs present in a blood sample. Blood samples were collected via venipuncture at the specified time frames. Week 0 corresponds to the last day of the treatment period in the parent study and Day 1 of the treatment period in the OLE study.
Time Frame: Week 0 (Week 0 = Day 1), Week 12, Week 24, Week 36, Week 48, Week 56
Population: OLE Safety Analysis Set: all participants who received at least 1 dose of daxdilimab in the OLE study. The overall number of participants analzyed represents the number of participants contributing data to any individual timepoint within the table.
Measure: Mean (Standard Deviation); unit: Percentage change in pDCs count
Arm/Group | Placebo/Daxdilimab 200 mg Q12W | Daxdilimab 200 mg Q4W in Parent Study | Daxdilimab 200 mg Q12W/Daxdilimab 200 mg Q12W
Number analyzed (Participants) | 47 | 57 | 51
Percentage change in pDCs count
  Week 0: number analyzed (Participants) | 24 | 32 | 30
  Week 0 | 70.59 (225.39) | -58.37 (36.19) | -30.40 (50.67)
  Week 12: number analyzed (Participants) | 23 | 36 | 33
  Week 12 | 1.33 (142.08) | 13.57 (158.14) | -21.25 (66.97)
  Week 24: number analyzed (Participants) | 22 | 33 | 29
  Week 24 | -14.39 (164.63) | -24.98 (79.85) | -19.86 (77.23)
  Week 36: number analyzed (Participants) | 12 | 12 | 15
  Week 36 | 13.64 (255.67) | -41.36 (41.29) | -51.11 (35.28)
  Week 48: number analyzed (Participants) | 8 | 5 | 6
  Week 48 | -49.47 (34.54) | -58.65 (43.33) | -4.44 (74.93)
  Week 56: number analyzed (Participants) | 3 | 2 | 3
  Week 56 | -75.22 (14.11) | -43.13 (49.49) | 4.15 (96.43)

6. Secondary Outcome: Number of Participants Expressing Anti-drug Antibodies (ADA)
Description: ADA incidence is the number of the participants with ADA positive post-Baseline only or boosted their preexisting ADA during the trial. Persistent positive was defined as ADA positive at ≥ 2 post-Baseline assessments (with ≥ 16 weeks between first and last positive) or positive at last post-Baseline assessment. Transient positive was defined as ADA post-Baseline positive but did not fulfill the criteria of persistent positive.
Time Frame: Up to approximately 56 weeks
Population: Any Daxdilimab Analysis Set: all participants who received at least 1 dose of daxdilimab in parent study or OLE study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Daxdilimab 200 mg Q12W | Daxdilimab 200 mg Q4W in Parent Study | Daxdilimab 200 mg Q12W/Daxdilimab 200 mg Q12W
Number analyzed (Participants) | 47 | 57 | 51
Participants
  ADA not detected | 34 | 48 | 44
  ADA Incidence | 7 | 6 | 4
  Only Baseline positive | 0 | 3 | 0
  Only post-Baseline positive | 6 | 3 | 3
  Both Baseline and post-Baseline positive | 7 | 3 | 2
  Persistent positive | 4 | 3 | 2
  Transient positive | 9 | 3 | 3

ADVERSE EVENTS:
Time Frame: Up to approximately 56 weeks
Description: Serious and other AEs is reported for the OLE Safety Analysis Set: all participants who received at least 1 dose of daxdilimab in the OLE study. All-cause mortality is reported for all participants enrolled/randomized in the study.
Arm/Group | Placebo/Daxdilimab 200 mg Q12W | Daxdilimab 200 mg Q4W in Parent Study | Daxdilimab 200 mg Q12W/Daxdilimab 200 mg Q12W
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/57 | 0/51
Serious Adverse Events (participants affected / at risk) | 3/47 | 5/57 | 5/51
Other Adverse Events (participants affected / at risk) | 12/47 | 19/57 | 19/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Daxdilimab 200 mg Q12W (N=47) | Daxdilimab 200 mg Q4W in Parent Study (N=57) | Daxdilimab 200 mg Q12W/Daxdilimab 200 mg Q12W (N=51)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus nephritis (Infections and infestations) | 0 | 1 | 0
Dengue fever (Infections and infestations) | 0 | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 1 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1
Glomerulonephritis minimal lesion (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Daxdilimab 200 mg Q12W (N=47) | Daxdilimab 200 mg Q4W in Parent Study (N=57) | Daxdilimab 200 mg Q12W/Daxdilimab 200 mg Q12W (N=51)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 3
COVID-19 (Infections and infestations) | 4 | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 3 | 1
Sinusitis (Infections and infestations) | 1 | 2 | 3
Urinary tract infection (Infections and infestations) | 1 | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1
Headache (Nervous system disorders) | 3 | 3 | 1
Depression (Psychiatric disorders) | 0 | 2 | 3
Insomnia (Psychiatric disorders) | 0 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4
Hypertension (Vascular disorders) | 4 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT05430854/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT05430854/SAP_001.pdf